CLINICAL TRIAL: NCT02917551
Title: Bacteremia Antibiotic Length Actually Needed for Clinical Effectiveness- BALANCE on the Wards: A Pilot RCT
Brief Title: BALANCE on the Wards: A Pilot RCT
Acronym: BALANCE-Wards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 218-2016
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Bacteremia
Keywords: Bacteremia, duration, non-critically ill, non-ICU
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shorter duration (7 days) (Active Comparator): Patients in 7 day arm will receive adequate antibiotics until the end of day 7 only
  Interventions: Other: 7 days of adequate antibiotic treatment
- Longer duration (14 days) (Active Comparator): Patients in 14 day arm will receive adequate antibiotics until the end of day 14 only
  Interventions: Other: 14 days of adequate antibiotic treatment

INTERVENTIONS:
Other: 7 days of adequate antibiotic treatment
  Arms: Shorter duration (7 days)
Other: 14 days of adequate antibiotic treatment
  Arms: Longer duration (14 days)

SUMMARY:
The burden of bloodstream infections is large and increasing over time. Antibiotic overuse continues to drive increased rates of antimicrobial-resistant pathogens across Canada. However, prospective audits have revealed that 30-50% of antibiotic utilization is unnecessary or inappropriate. If shorter duration therapy is as effective as longer duration therapy for these infections, antimicrobial consumption would be decreased. A pilot trial (approved by the Sunnybrook Research Ethics Board), is underway in critically ill patients at 17 Canadian ICUs. Investigators have successfully demonstrated feasibility with respect to protocol adherence and recruitment rates in the ICU. Investigators now aim to conduct a similar pilot RCT among non-ICU patients admitted to hospital wards with bloodstream infections to determine feasibility and protocol adherence of the same trial protocol.

DETAILED DESCRIPTION:
Bloodstream infections are a common and serious problem, and are associated with increased morbidity and mortality. At the same time, antibiotic overuse is also a common and serious problem, in that 30-50% of antibiotic use is unnecessary or inappropriate, and results in avoidable drug side effects such as kidney failure, Clostridium difficile infection, increased costs, and spiraling antibiotic resistance rates. The greatest contributor to antibiotic overuse is excessive durations of treatment.

Extensive research has demonstrated that shorter duration antibiotic treatment (less or equal to 7 days) is as effective as longer duration treatment for a variety of infectious diseases, but this question has not been directly studied in the setting of bloodstream infection. Our team's systematic review of the medical literature, national survey of Canadian infectious diseases and critical care physicians, and multicentre retrospective study all support the need for a randomized controlled trial comparing shorter (7 days) versus longer (14 days) antibiotic therapy for bloodstream infections.

Prior to performing the main trial, our pilot RCT in critically ill patients is near-completion.

In order to increase the generalizability to non-critically ill patients, Investigators want to conduct a similar pilot RCT in non-critically ill patients (BALANCE on the Wards) to establish the feasibility of the research design, and to optimize the definitive trial.

Investigators will conduct a randomized concealed allocation trial of shorter duration (7 days) versus longer duration (14 days) antibiotic treatment for patients with bloodstream infections across all non-ICU hospital wards in Sunnybrook Hospital (BALANCE on the Wards). Our ongoing BALANCE pilot RCT in ICU is approved by the Sunnybrook REB (PIN: 187-2014). The BALANCE on Wards pilot trial will use the same protocol, informed consent form and the case report forms that are approved by the Sunnybrook REB with minimal changes to make it ward specific. If the investigators are able to achieve the primary outcome of this trial in Sunnybrook hospital, the main BALANCE trial will potentially involve enrolment of non-ICU patients at all (or a subset of) participating sites.

If eligibility criteria and study procedures are substantially unchanged, results of the both the pilot BALANCE RCTs will be rolled into the dataset for the main BALANCE RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is in the hospital ward and not in the intensive care units at time the blood culture result reported as positive AND
2. Patient has a positive blood culture with pathogenic bacteria

Exclusion Criteria:

1. Patient already enrolled in either of the BALANCE trials
2. Patient is admitted in the ICU at the time of enrollment
3. Patient has severe immune system compromise, as defined by: absolute neutrophil count <0.5x109/L; or is receiving immunosuppressive treatment for solid organ or bone marrow or stem cell transplant
4. Patient has a prosthetic heart valve or synthetic endovascular graft
5. Patient has documented or suspicion of syndrome with well-defined requirement for prolonged treatment:

   i) infective endocarditis; ii) osteomyelitis/septic arthritis; iii) undrainable/undrained abscess; iv) unremovable/unremoved prosthetic-associated infection
6. Patient has a single positive blood culture with a common contaminant organism according to Clinical Laboratory & Standards Institute (CLSI) Guidelines: coagulase negative staphylococci; or Bacillus spp.; or Corynebacterium spp.; or propionobacterium spp.; or Aerococcus spp.; or Micrococcus spp.
7. Patient has a positive blood culture with Staphylococcus aureus.
8. Patient has a positive blood culture with Candida spp. or other fungal species.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Feasibility | 15 days
  defined by: (a) the adherence to treatment duration protocol (proportion of treatment courses); and (b) the rate of recruitment (enrolled per month). Investigators will consider enrolling patients in hospital wards for the BALANCE main trial if 90% of antibiotic treatment courses are within 7± 2 days in the shorter duration treatment arm or 14 ± 2 days in the longer duration treatment arm; and, if recruitment rates of at least 4 patients per 4 weeks is achieved.

SECONDARY OUTCOMES:
Hospital mortality rates | recorded as alive or dead at hospital discharge following index positive blood culture for an expected average of 4 weeks assesses upto one year.
90-day mortality rates | recorded as alive or dead at 90 days following index positive blood culture
Relapse rates of bacteremia | upto 30 days after adequate antibiotic treatment
  Defined as the recurrence of bacteremia due to original infecting organism (same Genus and species) after documentation of negative blood cultures or clinical improvement and within 30 days after completing course of adequate antimicrobial therapy.
Antibiotic allergy and adverse events | up to 30 days from start of antibiotic treatment.
Rates of C. difficile infection in hospital | Upto 30 days after index blood culture collection date
Rates of secondary nosocomial infection with antimicrobial resistant organisms in hospital | upto 30 days after index blood culture collection date
Hospital length of stay | for the duration of Hospital stay, expected for an average of 30 days assessed up to 1 year
Antibiotic free days | no. of days patient remained without antibiotics for up to 30 days post index blood culture collection date

CONTACTS AND LOCATIONS:
Overall Officials: Nick Daneman, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (6):
- Canada (6):
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - North York General Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daneman N, Rishu AH, Pinto R, Arabi Y, Belley-Cote EP, Cirone R, Downing M, Cook DJ, Hall R, McGuinness S, McIntyre L, Muscedere J, Parke R, Reynolds S, Rogers BA, Shehabi Y, Shin P, Whitlock R, Fowler RA; Canadian Critical Care Trials Group. A pilot randomized controlled trial of 7 versus 14 days of antibiotic treatment for bloodstream infection on non-intensive care versus intensive care wards. Trials. 2020 Jan 15;21(1):92. doi: 10.1186/s13063-019-4033-9. PMID 31941546